CLINICAL TRIAL: NCT05064774
Title: The Efficacy of Myofascial Release at the Cervicothoracic Region in Patients With Rotator Cuff Repairs: A Randomized Controlled Pilot Study
Brief Title: The Efficacy of Myofascial Release at the Cervicothoracic Region in Patients With Rotator Cuff Repairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sumeyye Cildan Uysal, MSc, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60116787-020/41785
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Rotator Cuff Tears
Keywords: myofascial release; rotator cuff tears; physiotherapy; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Myofascial Release Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomised controlled study this study was conducted with rotator cuff tear patients who underwent arthroscopic rotator cuff treatment.
  The patients' pain intensity, joint range of motion, flexibility of shoulder muscles, grip and muscle strength, shoulder function evaluations and physical characteristics, age, differences between body mass index were evaluated with Mann Whitney-U test.Measurements before and after treatment were evaluated with the Wilcoxon test. Friedman test was performed for the measurements made at postoperative 3, 7, and 12 weeks before in-group treatment. Bonferoni correction was done for possible differences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Patients who underwent arthroscopic rotator cuff repair surgery (n=10). They were implemented physiotherapy after the surgery once a week for 12 weeks. They were encouraged to do exercises 3 to 5 times every day.
  Interventions: Other: physiotherapy
- myofascial release group (Experimental): Patients who underwent arthroscopic rotator cuff repair surgery (n=10). They were implemented physiotherapy the same as the control group once a week for 12 weeks. In addition to physiotherapy they took myofascial release sessions twice a week for 4 weeks between 4 and 7 weeks.
  Interventions: Other: myofascial release technique; Other: physiotherapy

INTERVENTIONS:
Other: myofascial release technique — myofascial release group took myofascial release (MFR) therapy sessions twice a week for 4 weeks between 4 and 7 weeks. MFR was applied to upper trapezius, SCM, pectoralis major-minor and sternocostal fascia. muscle was replaced elongated position and pressure was applied for 60-120 second.
  Arms: myofascial release group
Other: physiotherapy — patients used sling up to 4 weeks. They did first 4 weeks passive/ assistive range of motion exercise. In 6-8 weeks they did active exercises. 8-12 weeks they did progressive resistive exercises.
  Other Names: classic physiotherapy

SUMMARY:
this study was conducted the patients with rotator cuff tears who underwent rotator cuff repair surger.The patients were randomly divided into 2 groups and a total of 20 subjects were randomized in a single block order using RandomAllocation Software 1.0.0 by simple randomization.All evaluation and treatment was done by the same physiotherapist.The first group was included in the traditional treatment program after rotator cuff repair, while the second group was included in the myofascial release program, 2 sessions a week between the 4th and 7th weeks, in addition to the traditional treatment.

DETAILED DESCRIPTION:
Patients in the 2 groups undergoing rc repair were also included in a similar physiotherapy program.Immobilization with a sling was made for 4-6 weeks after surgery. In addition to physiotherapy in group 2, myofascial release therapy was applied to the upper trapezius, sternocloidomastoideus, pectoral muscles (major, minor) 2 days a week between the 4th and 7th weeks after surgery, in addition to the conventional treatment. Myofascial treatment took 30-45 minutes per session.

ELIGIBILITY:
Inclusion Criteria:

* aged betweeen 18-65
* diagnosed with RC tear

Exclusion Criteria:

* wanting to leave the study
* not participating in assessments and/or treatments
* presence of massive tears
* accompanying nerve injuries,
* presence of labral lesion,
* diagnosed psychological problems,
* central nervous system problems
* those with any rheumatological and orthopedic diseases
* individuals who have had previous surgery on the same shoulder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
pain intensity | 12 weeks
  visual analog scale (pain during night, rest, activity), preoperative, post operative 3-7-12 weeks.
function | 12 weeks
  Constant Murley's score. This score has been used in preoperative, post operative 7-12 weeks. Higher score means better results. total point changes between 0-100.
quality of life ındex | 12 weeks
  short form-36 (SF-36) This scale is used in preoperative and pos operative 12 weeks.Higher score means better results.

SECONDARY OUTCOMES:
grip strength | 12 weeks
  Grip strength has been measured with dynamometer in preoperative, post operative 7-12 weeks.
flexibility | 12 weeks
  pectoralis minor flexibility was measured and saved as centimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeyye CILDAN UYSAL, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Page P. Shoulder muscle imbalance and subacromial impingement syndrome in overhead athletes. Int J Sports Phys Ther. 2011 Mar;6(1):51-8. PMID 21655457
- [Background] LeBauer A, Brtalik R, Stowe K. The effect of myofascial release (MFR) on an adult with idiopathic scoliosis. J Bodyw Mov Ther. 2008 Oct;12(4):356-63. doi: 10.1016/j.jbmt.2008.03.008. Epub 2008 Jun 4. PMID 19083694
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450